CLINICAL TRIAL: NCT01300806
Title: Impact of a Computer-Assisted SBIRT Program in an HIV Care Setting
Acronym: SBIRT
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 09035355
Record Dates: First submitted 2010-02-17; First posted 2011-02-23 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Substance Use
Keywords: HIV; harmful substance use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- myHERO SBIRT
- clinician administered SBIRT

SUMMARY:
The goal of this research is to assess the impact of the "screening, brief intervention, and referral to treatment" (SBIRT) intervention strategy for harmful substance use among HIV-positive people.

DETAILED DESCRIPTION:
The specific aims of the study are:

1. To assess the feasibility of conducting SBIRT using (1) a patient self-administered intervention embedded in a web-based Personal Health Record (PHR) compared to (2) a provider-administered SBIRT intervention guided by the Electronic Medical Record (EMR) during clinic appointments.
2. To examine the acceptability of web-based PHRs to conduct and communicate SBIRT compared to EMR-activated SBIRT conducted by clinic staff, from the perspective of the patient and the provider.
3. To assess the impact of SBIRT on risky drug and alcohol use in an HIV/AIDS population and subsequent effects on sexual risk behaviors and antiretroviral therapy (ART) adherence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* confirmed prior HIV+ serostatus
* ability to provide informed consent to be a participant over a 6 month period
* English or Spanish speaking

Exclusion Criteria:

Inability to answer questions with interviewer assistance. Not receiving primary care in clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic patients
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
reduced substance use among HIV-positive people | 6 months

SECONDARY OUTCOMES:
technological innovation to improve the quality of medical care | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol Dawson Rose, PhD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Derived] Dawson-Rose C, Draughon JE, Cuca Y, Zepf R, Huang E, Cooper BA, Lum PJ. Changes in Specific Substance Involvement Scores among SBIRT recipients in an HIV primary care setting. Addict Sci Clin Pract. 2017 Dec 12;12(1):34. doi: 10.1186/s13722-017-0101-1. PMID 29229000